CLINICAL TRIAL: NCT03328351
Title: Short-term Effect of Manual Therapy on Sensory Features in Patients With Cervical Radiculopathy: A Randomized Triple-blind Experimental Study
Brief Title: Effect of Manual Therapy on Sensory Features in Patients With Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dammam University
Record Dates: First submitted 2017-10-02; First posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Cervical Radiculopathy
Keywords: Manual therapy; cervical radiculopathy; pressure pain threshold; physiotherapy
MeSH Terms: conditions — Radiculopathy | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: triple-blind (The researcher was blinded to the outcome measures, whereas the assessor, who performed the outcome measures was blinded to the patient groups. The patient was blinded to treatment)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual group (Experimental): 1. The Manual therapy (Mobilization):
     1. Cervical postero-anterior vertebral mobilization glides: the mobilization was grade 3 for 2 min 3 set
     2. Cervical lateral vertebral glides: the mobilization was grade 3 for 1 min 3 set.
  2. Strengthening Exercises for deep neck flexor muscle
  Interventions: Other: manual therapy
- sham group (Sham Comparator): 1. Superficial soft tissue massage
  2. Strengthening Exercises: for deep neck flexor muscles for 10 seconds and repeating it for 10 times .
  Interventions: Other: Superficial soft tissue massage

INTERVENTIONS:
Other: manual therapy — 1. Manual therapy: One of the following techniques was used for the treatment group based on the patients' response (i.e centralization and reduction of symptoms).
     1. Cervical postero-anterior vertebral mobilization glides:
        a central posteranterior (PA) or unilateral PA oscillatory pressure of grade III on the patient's most symptomatic level for 2 minute and 3 sets .
     2. Cervical lateral vertebral glides :at grade III for 1 minute and 3 sets.
  2. Strengthening Exercises:
  for deep neck flexor muscles for 10 seconds and repeating it for 10 times.
  Other Names: mobilization; deep neck flexor exercise
  Arms: manual group
Other: Superficial soft tissue massage — 1. Superficial soft tissue massage: The researcher applied a superficial effleurage massage without moving the deeper tissue for 2 minutes for 3 sets
  Strengthening Exercises:
  for deep neck flexor muscles for 10 seconds and repeating it for 10 times
  Other Names: deep neck flexor exercise
  Arms: sham group

SUMMARY:
Background & Purpose: Cervical radiculopathy is a neurological disorder, which commonly results because of nerve compression. There are different types of physical therapy interventions that are used for cervical radiculopathy. The evidence of effectiveness of manual therapy in cervical radiculopathy is still limited. Short-term hypoalgesic effects after manual therapy was found in different musculoskeletal conditions. However, the effectiveness of manual therapy in patients with cervical radiculopathy hasn't been investigated yet. Therefore, the aim of study is to examine the short-term effect of manual therapy (mobilization) on the sensory features in patients with chronic cervical radiculopathy.

DETAILED DESCRIPTION:
Participants:

The sample size was calculated using G*power 3.1(F test, analysis of variance [ANOVA]: repeated measure, within between interaction, and a priori: compute required sample size). A result of 10 participants (treatment group=5 and sham group=5) was used to calculate the effect size (ES) of 0.44 for the pressure pain threshold on the cervical spine after the intervention(immediate effect) between group. The power estimated for ANOVA for the two group with a significance of 0.05 revealed that a total sample size of 28 participants was necessary to obtain a power of 0.80. . a minimum of 14 needed to be recruited in this study Participants with unilateral neck pain and radiating symptoms to upper extremity of more than three months were recruited from King Abdul-Aziz Hospital and East Jeddah general hospital in Jeddah, Saudia Arabia All patients signed a consent form before they participate in the study after explaining all procedures to them. The study was approved by the Institutional Review Board (IRB) at the University of Dammam (IRB Number: PGS-20160-30-142) and was approved by ministry of health at Saudia Arabia (IRB number: H-02J-002). All electronic data pertinent to the patients were being saved in a secured laptop, whereas the paper document will be kept in a locked cabinet.

Data analysis:

All statistical analysis was performed using IBM SPSS version 20 (Armonk, NY: IBM Corp). Significance levels will be set at p ≤ 0.05. Mean and standard deviation will be calculated as descriptive statistics. One-way repeated measures analysis of variance (ANOVA) and post hoc comparison, if needed will calculate the differences in the outcome measures: Quantitive sensory testing (QST), pain intensity, and active CROM

ELIGIBILITY:
Inclusion Criteria:

1. unilateral neck pain and radiating to upper extremity > 3 months.
2. age :between 35 to 65 years old.
3. Presence 3 out of 4 positive findings:

   * spurling test.
   * distraction test,
   * upper limb neurodynamic test for median nerve
   * ipsilateral cervical rotation test less than 60 degrees.

Exclusion Criteria:

1. osteoporosis.
2. tumor.
3. metabolic disease (DM,resting blood pressure are greater than 140/90).
4. rheumatoid arthritis.
5. history of whiplash injury.
6. myelopathy.
7. pregnancy.
8. history of cervical or thoracic surgery
9. generalized neurological disorders .
10. leg surgery or disease (fracture) -

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-12-18 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
pressure pain threshold (PPT) | Change from baseline in PPT at immediate post intervention
  An electronic algometer (Somedic AB, Farsta, Sweden) was used to quantify pain intensity (K pascal).
pressure pain threshold (PPT) | Change from baseline in PPT at 3 weeks post intervention
  An electronic algometer (Somedic AB, Farsta, Sweden) was used to quantify pain intensity (K pascal).

SECONDARY OUTCOMES:
Warmth/cold detection threshold and heat/cold pain threshold | Change from baseline in thermal detection & pain threshold at immediate post intervention
  A Thermotest System (SenseLab - Modular Sensory Analyser, Somedic AB, Horby, Sweden) was used to determine the thermal thresholds in degrees (°C )
Warmth/cold detection threshold and heat/cold pain threshold | Change from baseline in thermal detection & pain threshold at 3 weeks post intervention
  A Thermotest System (SenseLab - Modular Sensory Analyser, Somedic AB, Horby, Sweden) was used to determine the thermal thresholds in degrees (°C )
The Neck Disability Index (NDI) | Change from baseline in NDI at immediate post intervention
  The NDI is used to measure the patient reported disability in percentage
The Neck Disability Index (NDI) | Change from baseline in NDI at 3 weeks post intervention
  The NDI is used to measure the patient reported disability in percentage
Active Cervical Range of Motion | Change from baseline in CROM at immediate post intervention
  Cervical range of motion (CROM) device was used to assess the cervical range of motion in degree.
Active Cervical Range of Motion | Change from baseline in CROM at 3 weeks post intervention
  Cervical range of motion (CROM) device was used to assess the cervical range of motion in degree.
Numerical Pain Rating Scale (NPRS) | Change from baseline in NPRS at immediate post intervention
  The NPRS was used to assess a patient's level of pain in (11 points: 0 means no pain and 10 means severe pain.
Numerical Pain Rating Scale (NPRS) | Change from baseline in NPRS at 3 weeks post intervention
  The NPRS was used to assess a patient's level of pain in (11 points: 0 means no pain and 10 means severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ali M Alshami, PHD, Study Director — Imam Abdulrahman Bin Faisal University
Locations (2):
- Saudi Arabia (2):
  - East jeddah general hospital, Jeddah
  - king Abdulaziz hospital, Jeddah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alshami AM, Bamhair DA. Effect of manual therapy with exercise in patients with chronic cervical radiculopathy: a randomized clinical trial. Trials. 2021 Oct 18;22(1):716. doi: 10.1186/s13063-021-05690-y. PMID 34663421